CLINICAL TRIAL: NCT06222866
Title: Anticoagulation and Inflammation Monitoring in Patients After Heart and Vascular Interventions: Prospective Observational Study
Brief Title: Anticoagulation and Inflammation Monitoring in Patients After Heart and Vascular Interventions
Acronym: PAC-AIM
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: PAC-AIM
Record Dates: First submitted 2024-01-15; First posted 2024-01-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Heart Surgery; Vascular Surgery; Delirium; Hyperinflammatory Syndrome
Keywords: cardiac surgery; vascular surgery; Anticoagulation; Adverse Events; Monitoring; Delirium; Inflammation
MeSH Terms: conditions — Delirium; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after cardiovascular surgery who received anticoagulation: The investigated population comprises all patients after cardiovascular surgery who received anticoagulation. Subgroup analyses based on the level of inflammation, delirium, anticoagulation, and others will be conducted.
  Interventions: Diagnostic Test: Anticoagulation monitoring

INTERVENTIONS:
Diagnostic Test: Anticoagulation monitoring — Evaluation of different monitoring modalities to find the most appropriate anticoagulation monitoring tool for UFH therapy

SUMMARY:
The goal of this prospective observational study is to evaluate the most appropriate anticoagulation monitoring tool for unfractionated heparin (UFH), by comparison of different monitoring modalities in relation to adverse events occurrence (thrombosis/bleeding).

The main study questions are:

* What is the most appropriate anticoagulation monitoring tool (ACT, aPTT, viscoelastic tests (ROTEM), and anti-Xa) for UFH
* What is the incidence of adverse events associated with anticoagulation and inflammation after heart and vascular interventions
* Is there an association of available anticoagulation thresholds and monitoring tests with bleeding and/or thrombosis occurrence
* Is there an association of inflammation with delirium

Secondary study objectives include:

* Association of anticoagulation levels as measured by ACT, aPTT, viscoelastic tests (ROTEM), and anti-factor-Xa with adverse events
* Correlation of each anticoagulation monitoring test with the UFH anti-Xa measurement
* Correlation of each anticoagulation monitoring test with another (ACT, aPTT, ROTEM, anti-F-Xa) and the amount of blood loss post surgery
* The incidence of UFH-rebound effect and the need for protamine application
* Association of inflammation and increased / reduced need for anticoagulation titration
* Correlation of anticoagulation dosing with anticoagulation monitoring tests and adverse events
* The association of inflammation with adverse events
* The association and impact of inflammation on measured levels of anticoagulation with available tests
* Influence of anticoagulation on mortality
* Incidence of ECMO support
* Incidence of delirium (hypoactive and hyperactive) and correlation with vital (newly onset postoperative atrial fibrillation amongst others) and laboratory parameters, including, and pre-existing neurological disorders

DETAILED DESCRIPTION:
Patients undergoing major heart and vascular surgery are often in need of intraoperative and/or postoperative anticoagulation. To ensure the appropriate blood concentration of anticoagulants and reduce the risk of adverse events, anticoagulation monitoring is crucial. In contrast, due to contact of blood with artificial surfaces, some patients develop hyperinflammation which may increase the risk of thrombosis.

Patients undergoing heart surgery require full heparinization before the start of the heart-lung machine, which is later reversed using protamine. The levels of anticoagulation are intraoperatively monitored with activated clotting time (ACT). In the postoperative period, the monitoring of rest-heparinization or rebound effect is further performed. In certain cases, the addition of protamine is needed, based on the available monitoring tests. The postoperative monitoring of anticoagulation is usually performed using ACT and activated partial thromboplastin time (aPTT), and may be extended by other diagnostic methods, including viscoelastic tests. Moreover, to ensure the hemostatic capacity of the patient, monitoring of other parameters (platelet count, fibrinogen concentration, prothrombin time quick assay (PT), antithrombin level, etc.) may be included. Finally, in the case of patients receiving extracorporeal life support (ECMO), continuous anticoagulation is indicated, and its monitoring is of immense importance.

Furthermore, in the case of vascular surgery, patients require unfractionated heparin (UFH) intraoperatively, including postoperative continuous infusion.

The evidence on correlation and available monitoring tools is scarce and contradictory, usually based on retrospective analyses of patients´ data from medical charts. Additionally, the role of inflammation in the development of delirium is still unclear, and this association is a subject of debate.

Well-known consequences of postoperative delirium (POD) include poor functional outcome with increased morbidity and mortality, and increased healthcare costs due to institutionalization and rehospitalization. The incidence of POD after cardiac and vascular surgery remains between 13 and 52%. The current hypothesis on the pathophysiology of POD includes disruption of the blood-brain barrier allowing peripheral inflammation and mediators to cause neuro-inflammation. Neurotoxicity induced by a disbalance of pro- and anti-inflammatory mediators and oxidative stress might explain neuronal damage and neurotransmitter disbalance responsible for POD. To improve patients´ functional outcome and the financial burden of POD there is a growing interest in identifying predictive and diagnostic (bio-)markers. The neurofilament light chain (NfL) protein has shown promising results as a potential biomarker for POD. However, the literature on cardiac and vascular patients is limited.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 17 years
* Informed written consent
* Scheduled for cardiac intervention where the use of UFH is expected (elective surgery)
* Scheduled for vascular intervention when the need for perioperative anticoagulation is expected (elective surgery)
* Patients receiving ECMO support

Exclusion Criteria:

* Patients that are known to be pregnant
* Known participation in other interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients needing cardiac or vascular surgery who receive anticoagulation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events occurence | Patient follow-up of maximum 30 days
  Occurence of adverse events associated with anticoagulation monitoring and hyperinflammation

SECONDARY OUTCOMES:
ACT, aPTT, ROTEM, anti-factor Xa: Specific measured anticoagulation levels associated with adverse events | Patient follow-up of maximum 30 days
  Correlation and thresholds associated with adverse events
Correlation of each anticoagulation monitoring test with another (ACT, aPTT, ROTEM, anti-F-Xa) | Patient follow-up of maximum 30 days
  Correlation between various tests
Incidence of UFH-rebound and the need for protamine application | Patient follow-up of maximum 30 days
  The rate of UFH-rebound
Anticoagulation needs for patients receiving ECMO support and experiencing inflammation | Patient follow-up of maximum 30 days
  Anticoagulation range for patients with inflammation
Association of significant inflammation with adverse events | Patient follow-up of maximum 30 days
  Impact of inflammation on adverse events occurence
Incidence of ECMO support and delirium | Patient follow-up of maximum 30 days
  The rate of delirium, and the ECMO rate in patients after cardiovascular surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided
The decision will be made